CLINICAL TRIAL: NCT05728333
Title: Intravenous Adjuvant With Tirofiban Versus Alteplase Before Mechanical Thrombectomy in Acute Ischemic Stroke Patients With Large Vessel Occlusion: a Multicenter, Open Label, Randomized Controlled Trial.
Brief Title: Intravenous Tirofiban Versus Alteplase Before Mechanical Thrombectomy in Stroke
Acronym: ADJUVANT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADJUVANT
Record Dates: First submitted 2023-02-02; First posted 2023-02-15 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Acute Ischemic
Keywords: endovascular thrombectomy; large vessel occlusion; intravenous thrombolysis; tirofiban
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirofiban (Experimental): Tirofiban will be administrated intravenously before endovascular thrombectomy.
  Interventions: Drug: Tirofiban
- Alteplase (Active Comparator): Alteplase will be administrated intravenously before endovascular thrombectomy.
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Tirofiban — Intravenous tirofiban before endovascular thrombectomy.
  Other Names: Tirofiban & EVT
  Arms: Tirofiban
Drug: Alteplase — Intravenous alteplase before endovascular thrombectomy.
  Other Names: Alteplase & EVT
  Arms: Alteplase

SUMMARY:
In patients with acute ischemic stroke secondary to large vessel occlusion, the role of intravenous adjunctive medications, such as tirofiban, or alteplase before endovascular thrombectomy has not been well investigated. This trial aim to evaluate the efficacy and safety of intravenous tirofiban versus alteplase for acute ischemic stroke patients with large vessel occlusion piror to endovascular thrombectomy.

DETAILED DESCRIPTION:
Intravenous alteplase bridging with endovascular treatment (EVT) has been proven to be effective therapy in acute ischemic stroke patients due to large vessel occlusion (LVO). Several randomized controlled trials, aiming to explore the benefits and risks of intravenous alteplase prior to EVT in LVO stroke, have suggested that intravenous alteplase should not be omitted. Although intravenous alteplase results in successful reperfusion in approximately 10% to 20% of LVO patients, obviating the need for EVT, it has limitations. First, the time window for intravenous alteplase is narrow with strict indications and contraindications. Second, it may increase the risk of intracranial hemorrhage. Furthermore, alteplase is expensive. The above limitations lead to a very low proportion of patients who receive intravenous thrombolysis. Tirofiban is a selective IIb/IIIa receptor inhibitor, and it's effective in preventing thrombosis complications. Intravenous tirofiban has been increasingly used as an adjunctive treatment in acute ischemic stroke patients receiving EVT. However, a direct comparison between tirofiban and alteplase in LVO stroke has not been performed. We therefore conduct a randomized controlled trials to evaluate the efficacy and safety of intravenous tirofiban versus alteplase prior to EVT for acute ischemic stroke patients with LVO.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Presenting with acute ischemic stroke symptom.
3. Time from onset to hospital arrival:

   * (1) within 4.5 hours
   * (2) 4.5-9.0 hours, image inclusion criteria for the EXTEND trial must be met
   * (3) > 4.5 hours but within 24 hours, image inclusion criteria for the WAKE-UP trial must be met.
4. Eligible for intravenous thrombolysis.
5. Occlusion of the internal carotid artery, M1 or M2 segment of the middle cerebral artery, vertebrobasilar artery confirmed by CTA, MRA, or DSA.
6. Informed consent obtained from patients or their legal representatives.

Exclusion Criteria:

1. CT or MR evidence of hemorrhage (the presence of micro-bleeds is allowed);
2. Contraindications of IV rt-PA or tirofiban;
3. Contraindication to radiographic contrast agents, nickel, titanium metals or their alloys;
4. Arterial tortuosity and/or other arterial disease that would prevent the device from reaching the target vessel;
5. Patients with a preexisting neurological or psychiatric disease that would confound the neurological functional evaluations;
6. CT or MRI evidence of mass effect or intracranial tumor (except small eningioma);
7. CT or MRI evidence of cerebral vasculitis;
8. CTA or MRA evidence of intracranial arteriovenous malformations or aneurysms;
9. Any terminal illness with life expectancy less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional independence | 90 days post-endovascular treatment
  modified Rankin scale score of 0 to 2. (The modified Rankin scale scores range from 0 to 6, with 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

CONTACTS AND LOCATIONS:
Overall Officials: Congguo Yin, Doctor, Principal Investigator — Hangzhou First Hospital of Zhejiang University; Zhongming Qiu, Doctor, Principal Investigator — The 903rd Hospital of PLA, China
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the primary results was published

REFERENCES:
- [Result] Zi W, Qiu Z, Li F, Sang H, Wu D, Luo W, Liu S, Yuan J, Song J, Shi Z, Huang W, Zhang M, Liu W, Guo Z, Qiu T, Shi Q, Zhou P, Wang L, Fu X, Liu S, Yang S, Zhang S, Zhou Z, Huang X, Wang Y, Luo J, Bai Y, Zhang M, Wu Y, Zeng G, Wan Y, Wen C, Wen H, Ling W, Chen Z, Peng M, Ai Z, Guo F, Li H, Guo J, Guan H, Wang Z, Liu Y, Pu J, Wang Z, Liu H, Chen L, Huang J, Yang G, Gong Z, Shuai J, Nogueira RG, Yang Q; DEVT Trial Investigators. Effect of Endovascular Treatment Alone vs Intravenous Alteplase Plus Endovascular Treatment on Functional Independence in Patients With Acute Ischemic Stroke: The DEVT Randomized Clinical Trial. JAMA. 2021 Jan 19;325(3):234-243. doi: 10.1001/jama.2020.23523. PMID 33464335
- [Result] RESCUE BT Trial Investigators; Qiu Z, Li F, Sang H, Luo W, Liu S, Liu W, Guo Z, Li H, Sun D, Huang W, Zhang M, Zhang M, Dai W, Zhou P, Deng W, Zhou Z, Huang X, Lei B, Li J, Yuan Z, Song B, Miao J, Liu S, Jin Z, Zeng G, Zeng H, Yuan J, Wen C, Yu Y, Yuan G, Wu J, Long C, Luo J, Tian Z, Zheng C, Hu Z, Wang S, Wang T, Qi L, Li R, Wan Y, Ke Y, Wu Y, Zhu X, Kong W, Huang J, Peng D, Chang M, Ge H, Shi Z, Yan Z, Du J, Jin Y, Ju D, Huang C, Hong Y, Liu T, Zhao W, Wang J, Zheng B, Wang L, Liu S, Luo X, Luo S, Xu X, Hu J, Pu J, Chen S, Sun Y, Jiang S, Wei L, Fu X, Bai Y, Yang S, Hu W, Zhang G, Pan C, Zhang S, Wang Y, Cao W, Yang S, Zhang J, Guo F, Wen H, Zhang J, Song J, Yue C, Li L, Wu D, Tian Y, Yang J, Lu M, Saver JL, Nogueira RG, Zi W, Yang Q. Effect of Intravenous Tirofiban vs Placebo Before Endovascular Thrombectomy on Functional Outcomes in Large Vessel Occlusion Stroke: The RESCUE BT Randomized Clinical Trial. JAMA. 2022 Aug 9;328(6):543-553. doi: 10.1001/jama.2022.12584. PMID 35943471